CLINICAL TRIAL: NCT05620576
Title: Randomized, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate LY3857210 for the Treatment of Diabetic Peripheral Neuropathic Pain
Brief Title: A Chronic Pain Master Protocol (CPMP): A Study of LY3857210 in Participants With Diabetic Peripheral Neuropathic Pain (NP05).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18340; H0P-MC-NP05 (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 45 mg LY3857210 (Experimental): Participants received 45 milligram (mg) of LY3857210 orally once daily for up to 8 weeks.
  Interventions: Drug: LY3857210
- Placebo (Placebo Comparator): Participants received placebo orally once daily for up to 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3857210 — Administered orally
  Arms: 45 mg LY3857210
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This study is being done to test the safety and efficacy of the study drug LY3857210 for the treatment of diabetic peripheral neuropathic pain. This trial is part of the chronic pain master protocol H0P-MC-CPMP (NCT05986292) which is a protocol to accelerate the development of new treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have a visual analog scale (VAS) pain value greater than or equal to (≥) 40 and less than (<) 95 during screening.
* Have a history of daily pain for at least 12 weeks based on participant report or medical history.
* Have a body mass index <40 kilograms per meter squared (kg/m²) (inclusive).
* Are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain-relieving therapies (for example, physical therapy) and will not start any new nonpharmacologic pain-relieving therapies during study participation.
* Are willing to discontinue all pain medications taken for chronic pain conditions for the duration of the study.
* Have daily symmetrical foot pain secondary to peripheral neuropathy present for at least 6 months and as diagnosed through use of the Michigan Neuropathy Screening Instrument Part B ≥3 (©University of Michigan).
* Have a history and current diagnosis of type 1 or type 2 diabetes mellitus.
* Have stable glycemic control as indicated by a glycated hemoglobin less than or equal to (≤) 11 at time of screening.
* Are men, or women able to abide by reproductive and contraceptive requirements.

Exclusion Criteria:

* Have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest (for example, ablation techniques).
* Have surgery planned during the study for any reason, related or not to the disease state under evaluation.
* Have, in the judgment of the investigator, an acute, serious, or unstable medical condition or a history or presence of any other medical illness that would preclude study participation.
* Have substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5; American Psychiatric Association).
* Have had cancer within 2 years of baseline, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
* Have fibromyalgia.
* Are, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Have a positive human immunodeficiency virus (HIV) test result at screening.
* Have an intolerance to acetaminophen or paracetamol or any of its excipients.
* Have a history of alcohol, illicit drug, analgesic or narcotic use disorder within 2 years prior to screening.
* Have a current drug-induced neuropathy, for example, due to some types of chemotherapy, or other types of peripheral neuropathy.
* Have known hereditary motor, sensory or autonomic neuropathies.
* Have a seizure disorder, history of seizure (other than remote history of childhood febrile seizure), or a condition that would place the participant at increased risk of seizure, such as head injury (for example, skull fracture, cerebral contusion, concussion, or trauma resulting in prolonged. unconsciousness), intracranial neoplasm or hemorrhage.
* Are pregnant or breastfeeding.
* Have known or history of gastric or duodenal ulcers.
* Have known or history of inflammatory bowel disease (including ulcerative colitis or Crohn's disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (30):
- United States (28):
  - Synexus Clinical Research US, Inc., Chandler, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Accel Research Sites- Clinical Research Unit, DeLand, Florida
  - Suncoast Research Group, Miami, Florida
  - University of Miami Don Suffer Clinical Research Building, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research US, Inc - Orlando, Orlando, Florida
  - Synexus Clinical Research US, Inc., Pinellas Park, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Lillestol Research, Fargo, North Dakota
  - META Medical Research Institute, Dayton, Ohio
  - Altoona center for clinical research, Duncansville, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
  - Synexus Clinical Research - St. Petersburg, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Puerto Rico (2):
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Chronic Pain Master Protocol (CPMP): A Study of LY3857210 in Participants With Diabetic Peripheral Neuropathic Pain (NP05) — https://trials.lilly.com/en-US/trial/368106

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 45 mg LY3857210 | Placebo
Started | 87 | 44
Received at Least One Dose of Study Drug | 87 | 44
Completed | 80 | 37
Not Completed | 7 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Deviation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 45 mg LY3857210: Participants received 45 mg of LY3857210 orally once daily for up to 8 weeks.
- Total: Total of all reporting groups
Arm/Group | 45 mg LY3857210 | Placebo | Total
Number analyzed (Participants) | 87 | 44 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.7) | 63.7 (9.4) | 63.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 13 | 46
  Male | 54 | 31 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 19 | 61
  Not Hispanic or Latino | 45 | 25 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 75 | 38 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 44 | 131
Average Pain Intensity as Measured by the Numeric Rating Scale (NRS) [ [Mean (Standard Deviation); unit: score on a scale] — The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  score on a scale | 5.91 (1.58) | 5.62 (1.60) | 5.81 (1.59)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Pain Intensity as Measured by the Numeric Rating Scale (NRS)
Description: The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine.
  Posterior mean change from baseline, 95 percent (%) credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: All enrolled participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 45 mg LY3857210 | Placebo
Number analyzed (Participants) | 74 | 35
score on a scale | -1.70 [-2.11 to -1.30] | -1.81 [-2.40 to -1.21]
Statistical Analysis 1: Comparison: 45 mg LY3857210 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.10, 95% CI 2-sided [-0.61 to 0.82] — Posterior mean difference with 95% credible interval is reported

2. Secondary Outcome: Change From Baseline in the Brief Pain Inventory-Short Form Modified (BPI-SFM) Total Pain Interference Score
Description: The BPI-SFM is a numeric rating scale that assesses the severity of pain (severity scale) and its impact on daily functioning (Pain Interference scale). BPI-SFM pain interference scale has been reported here. Pain interference scale has 7 items, including general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life each assessed on a 10-point scale. All the 7-items are averaged to produce a total score ranging from 0 to 10 where, 0=does not interfere to 10=completely interferes and the mean is reported here. Higher score represents worse outcome. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 45 mg LY3857210 | Placebo
Number analyzed (Participants) | 77 | 36
score on a scale | -1.45 [-1.88 to -1.01] | -1.71 [-2.34 to -1.08]
Statistical Analysis 1: Comparison: 45 mg LY3857210 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.26, 95% CI 2-sided [-0.47 to 0.99] — Posterior mean difference with 95% credible interval is reported

3. Secondary Outcome: Change From Baseline in Overall Improvement as Measured by Patient's Global Impression of Change (PGIC)
Description: Patient's global impression of change captured the participant's perspective of treatment apart from sub-aspects of the general improvement. This is a numeric scale from 1 to 7: 1 = very much better, and 7 = very much worse.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 45 mg LY3857210 | Placebo
Number analyzed (Participants) | 78 | 36
score on a scale | 2.83 [2.58 to 3.08] | 2.51 [2.14 to 2.87]
Statistical Analysis 1: Comparison: 45 mg LY3857210 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.33, 95% CI 2-sided [-0.11 to 0.78] — Posterior mean difference with 95% credible interval is reported

4. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: The NRS was used to describe pain severity. Participants were asked to describe their worst pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 45 mg LY3857210 | Placebo
Number analyzed (Participants) | 74 | 35
score on a scale | -1.69 [-2.12 to -1.25] | -1.89 [-2.52 to -1.25]
Statistical Analysis 1: Comparison: 45 mg LY3857210 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.20, 95% CI 2-sided [-0.56 to 0.96] — Posterior mean difference with 95% credible interval is reported

5. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: VAS was a graphic, single-item scale where participants were asked to describe their pain intensity over the past week, on a scale of 0 to 100: 0 = no pain, and 100 = worst imaginable pain. Participants completed the VAS by placing a line perpendicular to the VAS line at a point that described their pain intensity.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 45 mg LY3857210 | Placebo
Number analyzed (Participants) | 78 | 36
score on a scale | -25.44 [-30.50 to -20.39] | -24.67 [-31.96 to -17.32]
Statistical Analysis 1: Comparison: 45 mg LY3857210 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.77, 95% CI 2-sided [-9.41 to 7.75] — Posterior mean difference with 95% credible interval is reported

6. Secondary Outcome: Change From Baseline on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale) - Average Hours of Sleep
Description: The MOS Sleep Scale consists of 12 questions addressing the past week. Question 1 asks time to fall asleep and it is reported in 5-point timeframe categories. Question 2 asks average hours of sleep. In the remaining 10 questions participants report how often a sleep symptom or problem was present on a scale ranging from '0=all of the time' to '5=none of the time.' MOS Sleep scale dimension scores range from 0 to 100 with lower score indicating improvement, except for the dimension of sleep adequacy, where higher scores indicate improvement. Here, the average hours of sleep (i.e., Question 2) is reported as the average number of hours slept each night during the past week (range 0 to 24 hours). Higher number of hours slept indicates improvement.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: hours per night
Arm/Group | 45 mg LY3857210 | Placebo
Number analyzed (Participants) | 78 | 36
hours per night | 0.07 [-0.15 to 0.30] | 0.21 [-0.11 to 0.53]
Statistical Analysis 1: Comparison: 45 mg LY3857210 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.13, 95% CI 2-sided [-0.51 to 0.24] — Posterior mean difference with 95% credible interval is reported

7. Secondary Outcome: Change From Baseline on the EuroQuality of Life Five Dimensions (5D) Five Level (5L) Questionnaire (EQ-5D-5L) Health State Index (United States Algorithm)
Description: The EQ-5D-5L assessed quality of life based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant was asked to 'check the ONE box that best describes your health TODAY,' choosing from 5 options (no problems, slight problems, moderate problems, severe problems, extreme problems) provided under each dimension. The scores in the 5 dimensions were summarized into a health state index score using the United States algorithm. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health: 0=a health state equivalent to death, and 1=perfect health.
  Posterior mean change from baseline, 95% credible intervals was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 45 mg LY3857210 | Placebo
Number analyzed (Participants) | 78 | 36
score on a scale | 0.06 [-0.01 to 0.12] | 0.07 [-0.02 to 0.15]
Statistical Analysis 1: Comparison: 45 mg LY3857210 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.01, 95% CI 2-sided [-0.11 to 0.08] — Posterior mean difference with 95% credible interval is reported

8. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Daily Dosage
Description: Total amount of rescue medication use as measured by average daily dosage. Posterior mean and 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milligram per day
Arm/Group | 45 mg LY3857210 | Placebo
Number analyzed (Participants) | 74 | 35
milligram per day | 156.82 [81.73 to 231.29] | 133.80 [28.09 to 240.77]
Statistical Analysis 1: Comparison: 45 mg LY3857210 vs Placebo; Test type: Superiority; Posterior Mean Difference = 23.02, 95% CI 2-sided [-108.05 to 152.33] — Posterior mean difference with 95% credible interval is reported

ADVERSE EVENTS:
Time Frame: Baseline through Week 8
Description: All enrolled participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- 45 mg LY3857210: Participants received 45 mg LY3857210 orally once daily for up to 8 weeks.
Arm/Group | 45 mg LY3857210 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/44
Serious Adverse Events (participants affected / at risk) | 2/87 | 1/44
Other Adverse Events (participants affected / at risk) | 16/87 | 7/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 45 mg LY3857210 (N=87) | Placebo (N=44)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 45 mg LY3857210 (N=87) | Placebo (N=44)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1/33 (1) | 0/13 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT05620576/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT05620576/SAP_001.pdf